CLINICAL TRIAL: NCT06892899
Title: Reducing the Burden of Post-traumatic Knee Osteoarthritis Targeting Persistent Abnormal Joint Loading and Quadriceps Muscle Dysfunctions in Young Adults With ACL Injury - a Pilot and Feasibility Study
Brief Title: Exercise Loading Biology Post-Traumatic OsteoArthritis Study - a Pilot and Feasibility Study
Acronym: ExeLoadBioPTOA
Status: Enrolling by invitation | Type: Observational
Sponsor: May Arna Risberg (Other)
Collaborators: Helse-Bergen HF (Other); Oslo University Hospital (Other)
Responsible Party: Sponsor-Investigator, May Arna Risberg, Professor, Norwegian School of Sport Sciences
Organization: Norwegian School of Sport Sciences (Other)
Other Study IDs: REK sør-øst C #644970
Record Dates: First submitted 2025-02-08; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2024-09

CONDITIONS: Anterior Cruciate Ligament Injury; Quadriceps Dysfunction; Knee Joint Loading; Anterior Cruciate Ligament Reconstruction; Risk Factors
Keywords: knee injury; anterior cruciate ligament injury; knee joint loading; quadriceps muscle strength; quadriceps muscle function; post-traumatic knee osteoarthritis; risk factors; prevention
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Knee Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Group 1: isolated injury: Group 2: combined injuries (concomitant injuries)

SUMMARY:
FROM RISK FACTORS TO THE PREVENTION OF LONG-TERM CONSEQUENCES AFTER CRUCIATE LIGAMENT INJURY (ACL injury) - This is a research project where we seek new knowledge about why some people have a high risk and others a low risk of developing long-term consequences such as persistent pain, thigh muscle dysfunctions and osteoarthritis after ACL surgery. Through more knowledge about risk factors for persistent pain, thigh muscle dysfunctions, and, in the long term, osteoarthritis, we have a greater opportunity to tailor preventive treatment measures to the individual.

We know that a subgroup of those who have undergone ACL surgery does not regain the normal function of the quadriceps muscle, that it does not become as strong as it used to or not quite the same as on the other healthy side. Some may notice this very well, others may not notice as much in the short term. We know that quadriceps dysfunctions can affect the biomechanical joint loading in your knee and can be a contributing risk factor to developing long-term consequences such as persistent pain, thigh muscle function and osteoarthritis after ACL injury.

We have methods to measure joint loading conditions in the knee and to identify changes in the cartilage, in the underlying bone tissue of the knee joint, and to measure various aspects of quadriceps muscle strength and dysfunctions.

In this study, we want to develop new knowledge about whether there is a difference in knee joint loading conditions and quadriceps muscle function between those who have low risk and those with a higher risk of developing post-traumatic osteoarthritis and whether there is an association between joint loading conditions in the knee after ACL surgery and quadriceps muscle function and symptoms.

DETAILED DESCRIPTION:
The main risk factors for knee OA disease are well-known: joint injuries and obesity. For those with ACL injury, systematic reviews have reported between 4 to 6 times increased risk of developing OA after ACL injury (PTOA). The following risk factors have been identified for PTOA in a recent systematic review by our OPTIKNEE group: ACL injury with concomitant injuries (meniscus and cartilage injuries), re-injuries after ACL injury, long-lasting quadriceps dysfunction, and inflammation after joint injury.

A better understanding of mechanisms to stratify the patients into different subgroups based on risk factors is critical. The mechanisms driving OA disease development are known to be 1) mechanical and 2) inflammatory. The mechanisms leading to PTOA combine mechanical, biological, structural, and neuromuscular factors.

Mechanical stress with persistent abnormal joint loading is an undisputed mechanism driving OA disease development. Altering joint mechanics (underloading and overloading) after ACL injury and reconstruction (ACLR) can lead to uneven stress and changes in stress across the articular cartilage of the joint surfaces, contributing to abnormal joint function and muscular dysfunction over time.

Whether such persistent abnormal knee joint loading patterns differ between individuals categorized as high risk compared to those at low risk of PTOA has not been investigated.

We do not understand the main drivers of the shifts in joint loading (underloading or overloading) or biochemical changes and whether this knowledge can be translated into developing joint-loading therapeutic interventions. However, we do know that quadriceps muscle weakness is a modifiable risk factor for non-traumatic OA and PTOA. ACL injury has shown a decline in quadriceps muscle function, which mimics ageing, known as sarcopenia. Quadriceps muscle dysfunction persists for some individuals for several years after ACLR, even after the cessation of structured rehabilitation, and has been questioned if it ever returns to normal. Despite decades of high-quality rehabilitation, normalizing quadriceps function in all ACL-injured and reconstructed patients remains unsolved.

This study has an overall aim of understanding more of the mechanisms for abnormal knee joint loading and quadriceps muscle dysfunctions in individuals at high- compared to low-risk PTOA (those with concomitant injuries and persistent symptoms compared to those with isolated ACL injury).

This cross-sectional study includes 40 participants 9 months to 2 years after ACLR with an extensive test-protocol of biomechanical-, neuromuscular- and biological assessments and tests. Hence, it is also a feasibility study for a planned randomized controlled trial of the effect of joint-loading therapeutic interventions on changes in knee joint loading for those at risk of developing PTOA. Furthermore, a sample of 40 individuals will be included to investigate primary outcomes' mean and standard deviation needed to calculate sample size for future randomized controlled trials.

Specific aims for the cross-sectional study are:

1. Investigate knee joint loading during gait, running and hopping, cellular, morphological, muscle inhibition and strength of the quadriceps muscle, and inflammatory knee joint markers in individuals who are 9 months to 2 years after an ACLR.
2. Characterize biomechanical, neuromuscular, and inflammatory factors in individuals classified as high-risk (concomitant injuries, persistent symptoms) for developing PTOA compared to those classified as low-risk (isolated ACL injury and no or minimal knee pain).
3. Explore the associations between abnormal knee joint loading, quadriceps muscle dysfunctions, and inflammatory markers in the knee joint 9 months to 2 years after ACLR
4. Describe the feasibility of the study regarding the recruitment of an extensive test-protocol
5. A pilot study for a future mechanistic RCT on the efficacy of a muscle- and joint-loading therapeutic exercise program on changes in knee joint loading and on surrogate outcomes of PTOA.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral ACL injury and ACLR (≤ one year between injury and surgery)

  * Surgery performed using the BPTB or hamstring grafts
  * Age between 16 and 40 years
  * Isolated ACL or with concomitant meniscal injury/cartilage injuries at surgery
  * Location (living) in the Oslo or Viken areas (due to the need for testing performed at the Norwegian School of Sport Sciences and Oslo University Hospital)
  * Healthy, uninjured contralateral knee

Exclusion Criteria:

* Above 40 years and below 16 years of age
* Previous ACL injury (re-rupture of graft or an ACL injury more than one year between injury and surgery)
* MCL/LCL grade 3 injuries
* Other lower extremity injuries less than one year before inclusion, or previous inflammatory arthropathy or systemic infection or inflammation
* Participants with bilateral ACL injuries

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants will be recruited through the Norwegian Knee Ligament Registry (NKLR). Established in 2004, its current data show that between 1800 and 2000 individuals go through ACL reconstruction annually in Norway. The NKLR includes nationwide data in Norway with >90% coverage for surgical data.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Tibiofemoral contact forces | The participant are tested once, as this is a cross-sectional study, 9 months to 2 years after ACLR
  Medial and lateral contact forces as a function of time during the standing phase of gait and the loading phase of running and hopping:
  * Walking and running over floor-embedded force plates (AMTI, Watertown, Massachusetts, USA)
  * Vertical and horizontal single-leg countermovement jumps with take-off and landing on a force platform.
  MSK modelling and Statistical Parametric Mapping (SPM) analysis will be used to provide a comprehensive understanding of the loading characteristics throughout the stance phase of gait and during the landing phases of each movement

SECONDARY OUTCOMES:
Patellofemoral contact forces | The participant are tested once, as this is a cross-sectional study, 9 months to 2 years after ACLR
  Walking, running and hopping - same as described for the Tibiofemoral contact forces.
Quadriceps and hamstring isokinetic muscle strength tests | The participant are tested once, as this is a cross-sectional study, 9 months to 2 years after ACLR
  Maximal Isokinetic leg extension and flexion strength in a dynamometer (HUMAC Norm, CSMi, Stoughton, MA, USA) at 60°/s
Leg press strength/power test | The participant are tested once, as this is a cross-sectional study, 9 months to 2 years after ACLR
  Seated leg press strength test: a Keiser Air300 horizontal pneumatic device with an A420 software (KeiserSport).
  The seat position is adjusted for each participant to result in approximately 90° of knee flexion. Participants will extend both legs with maximal effort for each repetition during the 10-repetition protocol. Maximum power and maximal force from the force-velocity profile of each leg will be used for further analysis
Voluntary quadriceps muscle activation test | The participant are tested once, as this is a cross-sectional study, 9 months to 2 years after ACLR
  The interpolated twitch technique (ITT) is used to evaluate voluntary muscle activation. Two percutaneous surface stimulation electrodes are placed over the distal and proximal parts of the quadriceps muscle belly

OTHER OUTCOMES:
Questionnaires including PROMs | The participant are tested once, as this is a cross-sectional study, 9 months to 2 years after ACLR
  The participants will out electronic questionnaires (Nettskjema; Sensitive Data (TSD), Oslo University). Participants characteristics, date of ACL injury/ diagnosis, date of ACLR, previous injuries or surgery, and re-injuries between surgery and inclusion are type of data to be answered. Furthermore, two validated patient-reported outcome measures (PROMs) the Knee Osteoarthritis Outcome Score (KOOS) subscales and the International Knee Documentation From (IKDC) are also included in the electronic questionnaires. All PROMs are scales from 0 (worst)-100 (best).
Magnetic Resonance Imaging (MRI) - bilateral | The participant are tested once, as this is a cross-sectional study, 9 months to 2 years after ACLR
  - The MRI Osteoarthritis Knee Score (MOAKS) (Hunter et al 2011) will be included as a semi-quantitative scoring method for different features in both knees scored from 0 (best) -4 (worst).
  The following quantified MRI sequences will also be included:
  * Fast spoiled gradient echo (FSPGR)
  * T2 and T2* mapping
  * Fat-supression T2mapping
Ultrasound (US) imaging of quadriceps | The participant are tested once, as this is a cross-sectional study, 9 months to 2 years after ACLR
  Muscle-architecture and 3D volume. US imaging data will be analyzed with specialized software 3D Slicer (3D Slicer image computing platform. (n.d.). 3D Slicer. Retrieved 3 February 2025, from https://slicer.org/) and Fiji (Schindelin et al. (2012). Fiji: An open-source platform for biological-image analysis. Nature Methods, 9(7), 676-682. https://doi.org/10.1038/nmeth.2019).
Biopsies of musculus vastus lateralis | The participant are tested once, as this is a cross-sectional study, 9 months to 2 years after ACLR
  Resting muscle biopsies will be obtained from the mid-portion of m. vastus lateralis from both legs. Biopsies are collected under local anesthesia (10 mg·ml-1 xylocaine + 5 µl·ml-1 adrenaline, AstraZeneca, London, UK) with a sterile 6-mm Bergstrom needle (Pelomi, Albertslund, Denmark). The main outcomes from the biopsy analyses will be compared to uninjured side: muscle fiber size for the different fiber types (e.g. Type I (slow) and Type II (fast)), fiber type distribution (description), satellite cells (description compared to uninjured side) and number of myonuclei, capillarization (description), and content of mitochondrial enzymes (description).
Synovial fluid samples | The participant are tested once, as this is a cross-sectional study, 9 months to 2 years after ACLR
  Synovial fluid will be collected by aspiration from the index joint with a 19G needle, using aseptic technique. Up to 10 ml will be aspirated (a minimum of 200 ul can be stored but aiming for at least 5 ml).
  Biomarkers: clinical markers (effusion grade, haemarthrosis grade) and synovial fluid molecular markers (candidate inflammatory markers IL-6 and MCP-1 as part of a limited panel of 'high risk' markers) for prediction of outcome, to compare in high- and low-risk groups. Grade of effusion in all participants attending face-to-face visits will be recorded prior to attempted aspiration (none/mild/moderate/large, using standard clinical grading), graded for blood content (none/mild/moderate/severe blood staining) as per published method and centrifuged at 3000G for 20 minutes at a controlled temperature of 20°C. The supernatants will be stored in cryovials at -80°C until use.
X-rays - bilateral | The participant are tested once, as this is a cross-sectional study, 9 months to 2 years after ACLR
  Radiographs (x-rays) will be taken utilizing a standardized protocol, weight-bearing, posterior-anterior radiographs, 10° caudal x-ray beam angulation with the use of a Synaflexer positioning frame. The x-rays will be scored based on the Osteoarthritis Research Society International (OARSI) scores and the Kellgren&Lawrence (KL) score from 0 (normal)- 4 (worst).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Sport Medicine, Norwegian School Sport Sciences, Oslo, Oslo County, Norway

IPD SHARING:
Plan to Share IPD: Undecided
As this is also a feasibility and pilot study. The PI, the co-PIs and the Scientific Advisory board will discuss this.